CLINICAL TRIAL: NCT03932786
Title: Research Into Visual Endpoints and RB Health Outcomes After Treatment (RIVERBOAT)
Brief Title: Studying Health Outcomes After Treatment in Patients With Retinoblastoma
Acronym: RIVERBOAT
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Debra Friedman, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC PED 1878; R01CA225005 (NIH); NCI-2019-00635 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2019-03-15; First posted 2019-05-01 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Retinoblastoma; Cancer Survivor; Biological Sibling; Intraocular Retinoblastoma; Unilateral Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue, saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective(biospecimens, vision assessment, questionnaires)
  Interventions: Procedure: Biospecimen collection; Other: Vision assessment; Other: Questionnaire administration; Other: Quality of life assessment; Other: Laboratory Biomarker Analysis
- Prospective (biospecimens, vision assessment, questionnaires)
  Interventions: Procedure: Biospecimen collection; Other: Vision assessment; Other: Questionnaire administration; Other: Quality of life assessment; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Biospecimen collection — Collection of tissue and saliva samples
Other: Vision assessment — Undergo vision assessment
Other: Questionnaire administration — Complete questionnaires
Other: Quality of life assessment — Complete questionnaires
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This trial studies health outcomes after treatment in patients with retinoblastoma. Gathering health information over time from patients and family members through vision assessments, samples of tissue and saliva, and questionnaires may help doctors learn more about what causes retinoblastoma, identify long-term health outcomes for patients with retinoblastoma, and find out which therapies may be the best for treating retinoblastoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define acute toxicity, subsequent malignant neoplasm (SMN) risk and visual outcomes in retinoblastoma (RB) survivors and compare patient centered psychosocial and neurocognitive and physical outcomes in survivors with normative data and sibling controls.

II. Create the first Clinically-Annotated Patient Tissues to Analyze Gene INteractions to assess biologic correlates of disease and facilitate future research: The RIVERBOAT-CAPTAIN biorepository, including germline deoxyribonucleic acid (DNA) and tumor tissue from patients, with detailed patient, disease and treatment-related information.

III. Using the RIVERBOAT-CAPTAIN clinically-annotated biorepository, determine the interplay between specific RB1 mutation type and the role of additional modifier genes in determining those tumor phenotypes that drive treatment decisions.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

RETROSPECTIVE COHORT: Patients treated between 2008-2018 undergo collection of saliva samples at >= 6 months after treatment, and undergo vision assessment at >= 6 months after treatment and again 1 year later if necessary. Previously collected tissue samples at the time of surgery are also obtained. Patients also complete questionnaires at >= 6 months after treatment and again 2 years later.

PROSPECTIVE COHORT: Patients treated between 2018-2023 undergo collection of saliva samples at the time of enrollment and at 6 months after treatment. Patients also undergo vision assessment at the time of enrollment, at 6 months, and 18 months after completion of treatment. Patients also complete questionnaires at 6 months and again 2 years later, as well as undergo collection of tissue samples at the time of surgery. Immediate family members with history of RB or RB1 gene mutation also undergo collection saliva samples.

ELIGIBILITY:
* Unilateral or bilateral intraocular retinoblastoma
* Diagnosis between the ages of 0 - 17.99 years
* Diagnosis on or after January 1, 2008
* No exclusions based on primary or secondary treatment modalities
* Retrospective group patients must be ≥ 6 months post end of treatment at study entry

  * For those already at this timepoint, they are now eligible
  * For those in treatment, or otherwise not yet at this timepoint, they are eligible once at they are ≥ 6 months post end of treatment
  * Prospective group patients must not have begun treatment
* Patients with diminished capacity will not be enrolled.
* Language: Patients must be able to communicate in English, French, or Spanish
* Sibling Cohort: One sibling, not affected by retinoblastoma will be enrolled, preference for the sibling closest in age to the RB patient.
* Regulatory Requirements: All patients and/or their parents or legal guardians must sign a written informed consent. All institutional, FDA, and NCI requirements for human studies must be met.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective patients (those treated between 2008 and 2018) identified by each site at the start of the study period and prospective patients (those treated between 2018 and 2023) identified at the time of diagnosis by each site during the study period with unilateral or bilateral intraocular retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute toxicity | Up to 1 year
Estimate malignant neoplasm (SMN) risk .Measured through medical record abstraction, | Up to 1 year
Assess visual outcomes measured via age appropriate visual acuity testing | Up to 1 year
Assess psycho-social outcomes utilizing questionnaires: BRIEF | Up to 2 years
Genes will be tested to examine the role they play in Retinoblastoma. This will be done via whole-exome sequencing and whole RB1 Gene examination. | Up to 1 year
Assess quality of life utilizing questionnaires: BRIEF | Up to 2 years
Assess quality of life utilizing questionnaires: CBCL | Up to 2 years
Assess quality of life utilizing questionnaires: Youth Self-Report | Up to 2 years
Assess quality of life utilizing questionnaires: Pediatric Quality of Life | Up to 2 years
Assess visual outcomes measured via parent report | Up to 1 year
Assess visual outcomes measured via vision questionnaires | Up to 1 year
Assess psycho-social outcomes utilizing questionnaires: BRIEF-P, | Up to 2 years
Assess psycho-social outcomes utilizing questionnaires: CBCL | Up to 2 years
Assess psycho-social outcomes utilizing questionnaires: Youth Self-Report | Up to 2 years
Assess psycho-social outcomes utilizing questionnaires: Pediatric Quality of Life | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Debra Friedman, MD, Principal Investigator — Vanderbilt Medical Center
Locations (11):
- United States (10):
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Illinois, Chicago, Chicago, Illinois
  - University of Minnesoa, Minneapolis, Minnesota
  - Washington School of Medicine at St. Louis, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Childeren's Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hosptial for Sick Children, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Undecided